CLINICAL TRIAL: NCT04163380
Title: Acute Effects of Resistance Training on Sex Hormone Concentrations on Different Phases of the Menstrual Cycle
Brief Title: Resistance Training and Sex Hormone Concentrations During the Menstrual Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Illinois University Edwardsville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 111B
Record Dates: First submitted 2019-10-30; First posted 2019-11-14 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-05

CONDITIONS: Women's Health
Keywords: Estrogen; Progesterone; Menstrual Cycle; Resistance Training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be blocked (four participants by block) and then randomized to start in one of the four menstrual cycle phases (EFP, LFP, ELP, or LLP). Their will be complete once they have gone through the four phases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early Follicular Phase (EFP) (Experimental)
  Interventions: Behavioral: Resistance Training
- Late Follicular Phase (LFP) (Experimental)
  Interventions: Behavioral: Resistance Training
- Early Luteal Phase (ELP) (Experimental)
  Interventions: Behavioral: Resistance Training
- Late Luteal Phase (LLP) (Experimental)
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — Participants will exercise at the mid-point of each menstrual cycle phase (EFP- day 4, LFP- day 11, ELP- day 18 and LLP- day 25 for a 28 day menstrual cycle). Training will consist of a warm up. Intensity will be set at 70% of 1RM, and the circuit training will include 7 strength exercises: leg press, rows, back squat, weighted crunches, deadlifts, bench press, and weighted squat jumps. The participant will perform 3 sets f 10 repetitions with 30 seconds of rest

SUMMARY:
Although there are numerous studies showing effects of aerobic training on sex hormone concentrations, research analyzing the fluctuation of sex hormones in response to resistance training (RT) is lacking. The objective of this project is to analyze estradiol (E2) and progesterone (P4) responses to an acute resistance training session throughout different phases of the menstrual cycle. This proposed research has strong implications for exercise prescription and for women in general, but more importantly will allow exercise physiologists, coaches, personal trainers, or nutritionists optimize exercise programming around women's menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Eumenorrheic females
* Age 18-45 years old
* BMI of 18.5-34.99 kg/m2

Exclusion Criteria:

* Practice exercise more than 2 days/week in the last 3 months.
* Cardiovascular, metabolic, pulmonary or muscular-skeletal condition
* Taking medications that affect metabolism (e.g. oral contraceptives)
* Irregular menstrual cycles

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 25 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in estrogen concentrations | through study completion, an average of 5 weeks
  Estrogen concentrations will be obtained from blood samples assessed using through ELISA kits
Change in progesterone concentrations | through study completion, an average of 5 weeks
  Progesterone concentrations will be obtained from blood samples assessed using through ELISA kits

SECONDARY OUTCOMES:
Lean body mass (kg) | At baseline: 1 assessment point
  Lean body mass (kg) will be assessed through Dual-energy X-ray Absorptiometry
Fat mass (kg) | At baseline: 1 assessment point
  Fat mass (kg) will be assessed through Dual-energy X-ray Absorptiometry
Relative body fat (%) | At baseline: 1 assessment point
  Relative body fat (%) will be assessed through Dual-energy X-ray Absorptiometry
Skeletal muscle mass (kg) | At baseline: 1 assessment point
  Skeletal muscle mass (kg) will be estimated using Dual-energy X-ray Absorptiometry values
Cardiorespiratory Fitness | At baseline: 1 assessment point
  Cardiorespiratory Fitness will be assessed with a cardiopulmonary exercise test using the Bruce protocol
Strength in Bench Press | At baseline: 1 assessment point
  Maximal strength bench press will be assessed using one repetition maximum test
Strength in Leg Press | At baseline: 1 assessment point
  Maximal strength in leg press will be assessed using one repetition maximum test
Changes in diet | through study completion, an average of 5 weeks
  Diet will be assessed using the a 24h dietary recall

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Illinois University Edwardsville, Edwardsville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No